CLINICAL TRIAL: NCT06470035
Title: A Randomized, Double Blind Sham Controlled Clinical Trial to Evaluate the Efficacy of Electrical Vestibular Nerve Stimulation (VeNS), Compared to a Sham Control for Treatment of Major Depressive Disorder (MDD) - Modius Mood Study
Brief Title: Electrical Vestibular Nerve Stimulation (VeNS) as a Treatment for Major Depressive Disorder (MDD)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neurovalens Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MMS002
Record Dates: First submitted 2024-06-14; First posted 2024-06-24 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Major Depressive Disorder (MDD; Depressive Disorder, Major
Keywords: VeNS; Depression; MDD; Vestibular stimulation
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active VeNS (Experimental): The active device utilizes a technology termed vestibular nerve stimulation (VeNS). The device will be placed on the head in a manner analogous to headphones and will deliver a small electrical current to the skin behind the ears, over the mastoid processes. Participants will be advised to use the device at home for 30 minutes per day.
  Interventions: Device: Active VeNS Device
- Sham VeNS (Sham Comparator): The sham device looks identical to the active device and interacts with the app in a similar manner to the active device. The device will be placed on the head in a manner analogous to headphones with hydrogel electrodes placed over the mastoid processes. Participants will be advised to use the device at home for 30 minutes per day.
  Interventions: Device: Sham VeNS Device

INTERVENTIONS:
Device: Active VeNS Device — Battery powered non-invasive neurostimulation device
  Other Names: Modius Mood
  Arms: Active VeNS
Device: Sham VeNS Device — Placebo comparator sham device (no active stimulation)
  Arms: Sham VeNS

SUMMARY:
Trial title: A Randomized, Double Blind Sham Controlled Clinical Trial to Evaluate the Efficacy of Electrical Vestibular Nerve Stimulation (VeNS), Compared to a Sham Control for Treatment of Major Depressive Disorder (MDD) - Modius Mood Study

The aim of this study: To better evaluate the efficacy of non-invasive electrical vestibular nerve stimulation (VeNS) as a method of treating major depressive disorder(MDD) , as compared to a sham control.

Allocation: Randomized to either active device or control device usage.

Endpoint classification: Efficacy Study Intervention Model: Parallel Assignment in 1:1 active to control allocation

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent
2. Adults, (US ≥ 22 years and ≤ 80 years, UK ≥ 18 years and ≤ 80 years) male or female at the time of signing informed consent
3. Beck's Depression Inventory-ll (BDI-ll) score of ≥ 14 at Screening
4. Established diagnosis of depression as confirmed at the time of screening by the Mini-International Neuropsychiatric Interview (MINI)
5. A Generalized Anxiety Disorder (GAD-7) score <10 at screening
6. On anti-depressant medication to treat depression (participant must only be on one Selective Serotonin or Norepinephrine Reuptake Inhibitor (SSRI/SNRI) for at least 1 year prior to baseline visit, and no longer than 5 years)
7. Stable dose of current prescribed antidepressant (SSRI/SNRI) medication to treat depression, 3 months prior to baseline appointment
8. Maintain a stable prescribed medication and/or treatment regime to treat depression for the duration of the trial
9. No change in regular medication for the duration of the trial (unless directed by a health care provider).
10. Can speak / read English
11. Ability and willingness to complete all study visits and procedures; in particular an agreement to engage with trying to use the device per the study protocol
12. Ability and willingness to adhere to 30 minutes usage of the device daily for the duration of the trial
13. Access to Wi-Fi for the duration of the study
14. Access to a computer, laptop, iPad, tablet or smartphone (to complete study visits and complete online study questionnaires)
15. Willingness to use a video calling platform to conduct remote study visits
16. Agree not to undergo any extreme lifestyle changes during the duration of the study that could impact mood e.g. dietary , exercise changes
17. Agree not to begin any complimentary or alternative therapies that may affect your mood during the time on the study e.g use of mental health apps, CBT

Exclusion Criteria:

1. Risk of persistent self-harm or suicide as confirmed by the Columbia Suicide Severity Rating Scale (CSSRS)
2. Diagnosis or history of bipolar disorder
3. History of or a current psychotic disorder such as schizophrenia or other non-mood disorder psychosis
4. Diagnosis of substance use disorder within the past 12 months or current substance use dependence
5. Use of recreational drugs (e.g nalgesics, depressants, stimulants, and hallucinogens). Subject can enrol after a washout period of 30 days
6. Female who is pregnant or breast-feeding
7. History of diagnosed cognitive impairment / disorder such as delirium or dementia
8. Previous or current diagnosis of a chronic viral infection, for example hepatitis or HIV (potential damage to vestibular system, known as vestibular neuropathy).
9. History of stroke or head injury requiring intensive care or neurosurgery (potential damage to neurological pathways affected by vestibular stimulation)
10. Presence of permanently implanted batterypowered medical device or stimulator (e.g., pacemaker, implanted defibrillator, deep brain stimulator, vagal nerve stimulator, etc.)
11. History of epilepsy
12. History of severe tinnitus or vertigo
13. History of skin breakdown, eczema or other dermatological condition (e.g. psoriasis) affecting the skin behind the ears.
14. History or presence of malignancy within the last year (except basal and squamous cell skin cancer and in-situ carcinomas)
15. History of vestibular dysfunction or another inner ear disease
16. Regular use (more than twice a month) of antihistamine medication within the last 6 months. The subject can opt to switch to Fexofenadine (non-drowsy) and may enrol after a wash-out period of 2 weeks
17. Diagnosis of active migraines
18. Previous use of Modius device or any VeNS device
19. Participation in other clinical trials sponsored by Neurovalens
20. Participation in any other depression studies at the time of enrolment and throughout this study duration
21. Any other medical condition, or medication use, that in the opinion of the PI is likely to make the subject refractory to VeNS.
22. Failure to use device daily during trial participation (no more than 14 consecutive days usage drop without reasonable explanation)
23. Persistent failure to comply with study protocol and procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HDRS-17) | Change in score from baseline to 6 weeks
  The HDRS (also known as the HAM-D) is the most widely used clinician-administered depression assessment scale. The original version contains 17 items (HDRS-17) pertaining to symptoms of depression experienced over the past week. Scoring is based on the 17-item scale and scores of 0-7 are considered as being normal, 8-16 suggest mild depression, 17-23 moderate depression and scores over 24 are indicative of severe depression; the maximum score being 52 on the 17-point scale. The HDRS-17 scoring shall be the Primary Outcome of the study and will be completed at baseline and each study visit.
Hamilton Depression Rating Scale (HDRS-17) | 6 weeks
  The HDRS (also known as the HAM-D) is the most widely used clinician-administered depression assessment scale. The original version contains 17 items (HDRS-17) pertaining to symptoms of depression experienced over the past week. Scoring is based on the 17-item scale and scores of 0-7 are considered as being normal, 8-16 suggest mild depression, 17-23 moderate depression and scores over 24 are indicative of severe depression; the maximum score being 52 on the 17-point scale. The HDRS-17 scoring shall be the Primary Outcome of the study and will be completed at baseline and each study visit. The proportion (%) of participants achieving the HDRS-17 minimal clinically important difference (≥3 point reduction) by the 6-week time point between the active and sham groups.

SECONDARY OUTCOMES:
WHO Disability Assessment Schedule 2.0 (WHODAS2) | Change in score from baseline to 6 weeks
  The WHO Disability Assessment Schedule 2.0 is a standardized assessment tool developed by the World Health Organization (WHO) to measure general health, disability levels and impairment across various domains of functioning, including mental and neurological disorders. It is designed to assess the impact of health conditions and disabilities on an individual's ability to participate in various life activities. The WHODAS 2.0 shall be a secondary outcome of this study, and will be completed at the baseline visit and repeated at each visit.
Insomnia Severity Index (ISI) | Change in score from baseline to 6 weeks
  The Insomnia Severity Index (ISI) is a validated short, self-report screening assessment tool designed to evaluate insomnia by measuring an individual's perception of both day and night symptoms of insomnia. The Index consists of seven items which are each assessed in terms of perceived difficulty: falling sleep, staying asleep, and time of awakening, satisfaction with current sleep pattern, interference with daily functioning, noticeability by others of impact of lack of sleep, and degree of perceived distress or concern caused by the sleep problem. The ISI shall be a secondary outcome of the study and be completed at baseline and 6 weeks.
Quality of Life (EQ-5D-5L) | Change in score from baseline to 6 weeks
  The EQ-5D-5L is a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each level is rated on scale that describes the degree of problems in that area. The tool also has an overall health scale where the rater selects a number between 1-100 to describe the condition of their health, 100 being the best imaginable. The EQ-5L-5D shall be completed at baseline and at 6 weeks. The EQ-5L-5D has previously been tested for reliability and validity.
Hamilton Depression Rating Scale (HDRS-17) | Change in score at 4 week post-intervention timepoint
  The HDRS (also known as the HAM-D) is the most widely used clinician-administered depression assessment scale. The original version contains 17 items (HDRS-17) pertaining to symptoms of depression experienced over the past week. Scoring is based on the 17-item scale and scores of 0-7 are considered as being normal, 8-16 suggest mild depression, 17-23 moderate depression and scores over 24 are indicative of severe depression; the maximum score being 52 on the 17-point scale.
WHO Disability Assessment Schedule 2.0 (WHODAS2) | Change in score at 4 week post-intervention timepoint
  The WHO Disability Assessment Schedule 2.0 is a standardized assessment tool developed by the World Health Organization (WHO) to measure general health, disability levels and impairment across various domains of functioning, including mental and neurological disorders. It is designed to assess the impact of health conditions and disabilities on an individual's ability to participate in various life activities. The WHODAS 2.0 shall be a secondary outcome of this study, and will be completed at the baseline visit and repeated at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Peter Colvonen, Principal Investigator — San Diego Healthcare System
Locations (2):
- VA San Diego Healthcare System, San Diego, California, United States
- Biomedical Science Research University of Ulster, Coleraine, Belfast, Co.Antrim, United Kingdom

IPD SHARING:
Plan to Share IPD: No